CLINICAL TRIAL: NCT05507216
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Study to Evaluate the Efficacy and Safety of ABX464 Once Daily for Induction Treatment in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: ABTECT-2 - ABX464 Treatment Evaluation for Ulcerative Colitis Therapy -2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABX464-106
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABX464 50mg (Experimental): Subjects will be orally dosed daily in a fed condition (ideally at the same time in the morning) for 8 weeks
  Interventions: Drug: ABX464
- ABX464 25mg (Experimental): Subjects will be orally dosed daily in a fed condition (ideally at the same time in the morning) for 8 weeks
  Interventions: Drug: ABX464
- Placebo (Placebo Comparator): Subjects will be orally dosed daily in a fed condition (ideally at the same time in the morning) for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX464 — Administered once daily in the morning with food
  Other Names: Obefazimod
  Arms: ABX464 25mg; ABX464 50mg
Drug: Placebo — Administered once daily in the morning with food
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, placebo controlled study to evaluate the efficacy and safety of ABX464 given at 25 or 50 mg QD in inducing clinical remission in subjects with moderately to severely active ulcerative colitis who have inadequate response, no response, a loss of response, or an intolerance to either conventional therapies [corticosteroids, immunosuppressant (i.e. azathioprine, 6-mercaptopurine, methotrexate)] and/or advanced therapies [biologics (TNF inhibitors, anti-integrins, anti-IL-23), and/or S1P receptor modulators, and/or JAK inhibitors].

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 16 years old; Adolescent subjects will only be enrolled if approved by the country regulatory/health authority. If these approvals have not been granted, only subjects ≥ 18 years old will be enrolled. To be eligible, adolescent subjects must weigh ≥ 40 kg and meet the definition of Tanner Stage 5 at the screening visit.
* Subjects must understand, sign and date the written voluntary informed consent form at the visit prior to any protocol-specific procedures. For under-aged subjects, national requirements regarding consent should also be met.
* Documented diagnosis of UC confirmed by endoscopy and histology. Should endoscopy/histology results not be available at screening, results from endoscopies and biopsies taken at screening may be used.
* Active disease defined by modified Mayo score (MMS) ≥ 5 with rectal bleeding subscore (RBS) ≥ 1 and endoscopy subscore (MES) of 2 or 3 (confirmed by central reader).
* Subjects with documented inadequate response (defined as lack of response or loss of response or intolerance) to at least one of the following treatments: corticosteroids, immunosuppressant, biologic or biosimilar therapies, S1P receptor modulators and/or JAK inhibitors and/or new drugs approved during the study (note: failure to only 5-ASA or sulfasalazine is not accepted).
* Women of childbearing potential (WOCBP) subjects and male subjects with WOCBP partner must agree to comply with the contraception requirements described in the protocol.
* Subjects able and willing to comply with study visits and procedures as per protocol.
* Subjects should be affiliated to a health insurance policy whenever required by a participating country or state.

Exclusion Criteria:

* Subjects with UC limited to an isolated proctitis (≤ 15cm from anal verge) determined by endoscopy central reading.
* Subjects with primary sclerosing cholangitis or autoimmune hepatitis.
* Subjects who have failed on 5-ASA or sulfasalazine therapy only.
* Subjects with CD or presence or history of fistula, indeterminate colitis, infectious/ischemic colitis or microscopic colitis (lymphocytic and collagenous colitis).
* History or current evidence of toxic megacolon, fulminant colitis, bowel perforation.
* History of colonic cancer or colonic low grade or high grade dysplasia adenomatous polyps, and/or at the screening endoscopy, evidence of colonic cancer or evidence of low grade or high grade dysplasia adenomatous polyps (fully removed or not).
* Recent or planned bowel surgery or history of proctocolectomy or partial colectomy or current stoma.
* Subjects on antidiarrheals including those working on motility (e.g., loperamide, diphenoxylate with atropine, etc.).
* Subjects on probiotics (e.g., Culturelle® [Lactobacillus GG, i-Health, Inc.], Saccharomyces boulardii).
* Subjects who do not meet the washout period requirements prior to the screening endoscopy.
* Subjects with the following hematological and biochemical laboratory parameters obtained during the screening period:

  * Hemoglobin ≤ 8.0 g dL-1
  * Absolute neutrophil count < 750 mm-3
  * Platelets < 100,000 mm-3
  * Creatinine clearance < 60 mL.min-1 (Cockroft-Gault formula)
  * Total serum bilirubin > 1.5 x ULN
  * Alkaline phosphatase, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2 x ULN
* Subjects with the following conditions (infection):

  * Subjects with chronic or recurrent grade 3 or grade 4 infection within the last 2 months prior to screening or a history of opportunistic infection while not on immunosuppressive therapy.
  * Herpes zoster reactivation within the last 2 months prior to screening.
  * Subjects with active infection at screening or any major episode of infection that required hospitalization or treatment with intravenous antibiotics within 1 month of screening or during screening. Fungal infection of nail beds is allowed.
  * Positive assay or stool culture for pathogens (ova and parasite examination, bacteria) or positive test for Clostridium difficile toxin at screening. If C. difficile is positive, subject may be treated and retested ≥ 2 weeks after completing treatment.
  * Subjects with HIV infection.
  * Subjects having acute or chronic hepatitis B infection at screening (positive for hepatitis B surface antigen [HbsAg], or negative for HbsAg and positive for anti-hepatitis B core antibody in conjunction with detectable HBV DNA, or detectable HBV DNA).
  * Subjects having acute or chronic hepatitis C infection at screening as defined by positive for hepatitis C antibody (subjects successfully treated and without recurrence ≥ 1 year with no detectable HCV RNA [assessed centrally] are eligible).
  * Active tuberculosis (TB) or untreated latent TB are ruled out. For subjects with positive or intermediate QuantiFERON test see the current study protocol.
* Subjects with an uncontrolled ischemic heart disease and/or a history of congestive heart failure with New York Heart Association (NYHA) class 3 or 4 symptoms.
* Subjects with a family or personal history of congenital or acquired long QT syndrome, or subjects with a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval [Fridericia or Bazett correction] >450 milliseconds for male and > 460 milliseconds for female).
* Subjects with a history of torsade de pointe (TdP).
* Acute or chronic of clinically relevant pulmonary, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable central nervous system pathology such as seizure disorder, or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history (note: treated autoimmune hypothyroidy and autoimmune diabetes are allowed).
* Serious illness requiring hospitalization within 4 weeks prior to screening (except UC flare).
* Subjects previously treated with ABX464.
* Subjects with a known hypersensitivity to the active substance or to any of the excipients.
* WOCBP subject who is pregnant or breast-feeding at screening, or intends to become pregnant during the study, or male subject with WOCBP partner who intends to be pregnant during the study.
* Illicit drug or alcohol abuse or dependence.
* Subjects who received live vaccine within 3 months prior to screening and/or who's planning to receive such a vaccine during the study duration.
* Use of any investigational or non-registered product within 3 months or within 5 half-lives preceding baseline, whichever is longer, and during the study.
* Subjects committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
* Any condition, which in the opinion of the investigator, could compromise the subject's safety or adherence to the study protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve clinical remission per Modified Mayo Score at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on clinical remission

SECONDARY OUTCOMES:
Proportion of subjects who achieve endoscopic improvement at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on endoscopic improvement
Proportion of subjects who achieve clinical response per MMS at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on clinical response as per MMS
Proportion of subjects with symptomatic remission at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on symptomatic remission
Proportion of subjects with HEMI per Geboes at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on histologic-endoscopic mucosal improvement (HEMI)

CONTACTS AND LOCATIONS:
Overall Officials: Severine Vermeire, MD, PhD, Principal Investigator — UZ Leuven, Belgium; Bruce Sands, MD, PhD, Principal Investigator — Mount Sinai Health System Digestive Disease Institute, New York USA
Locations (273):
- United States (61):
  - University of Alabama -Birmingham, Birmingham, Alabama
  - Research Solutions of Arizona, PC, Litchfield Park, Arizona
  - Valleywise Health Medical Center, Phoenix, Arizona
  - Reliance Research, Scottsdale, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - National Institute of Clinical Research, Bakersfield, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Citrus Valley Gastroenterology, Covina, California
  - United Medical Doctors, Murrieta, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Clinical Applications Laboratories, San Diego, California
  - Kaiser Foundation Research Institute, a Division of Kaiser Permanente Hospitals, Aurora, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Superior Associates in Research, Hialeah, Florida
  - IHS Health, Kissimmee, Florida
  - Infinite Clinical Research Inc, Miami, Florida
  - Research Associates of South Florida, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Reliant Medical Research, LLC, Miami, Florida
  - Ocala GI Research, Ocala, Florida
  - Sarkis Clinical Trials - Parent, Ocala, Florida
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Alliance Clinical Research, Tampa, Florida
  - Iowa Digestive Disease Center, Clive, Iowa
  - The University of Iowa, Iowa City, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Gastrointestinal Associates, PA, Flowood, Mississippi
  - BVL Clinical Research, Liberty, Missouri
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - NY Scientific Corp., Brooklyn, New York
  - Mount Sinai, New York, New York
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Board of Regents of the University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Rapid City Medical Center, LLC, Rapid City, South Dakota
  - Digestive Health Research, LC, Hermitage, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Inquest Clinical Research, Baytown, Texas
  - Valley Institute of Research, Fort Worth, Texas
  - Mt.Olympus Medical Research, Katy, Texas
  - Digestive System Healthcare, Pasadena, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Gastroenterology Consultants and Endoscopy Center of Southwest Virginia, Roanoke, Virginia
  - The Vancouver Clinic, Vancouver, Washington
- Argentina (5):
  - CEMIC, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Centro de Investigacion CICE, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Gastroenterología Diagnóstica y Terapéutica (Gedyt), Ciudad Autonoma Buenos Aires
- Belgium (5):
  - GZA Ziekenhuizen, Antwerp
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Delta, Roeselare
- Brazil (15):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - Hospital Aliança, Salvador, Estado de Bahia
  - L2IP - Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - CDC - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Instituto de Pesquisas em Saúde - Fundação Universidade de Caxias do Sul (IPS/FUCS), Caxias do Sul, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - CECIP - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Pesquisare Saúde, Santo André, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - Irmandade da Santa Casa da Misericórdia de Santos, Santos, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC, São Bernardo do Campo, São Paulo
  - Hepatogastro, São Paulo, São Paulo
- Bulgaria (3):
  - DCC 'Sv. Pantaleymon' OOD, Pleven
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - MC Medica Plus, Veliko Tarnovo
- Canada (3):
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hopital Maisonneuve-Rosemont d/b/a CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
- Croatia (5):
  - General Hospital "Dr.Tomislav Bardek" Koprivnica, Koprivnica
  - Poliklinika Borzan d.o.o, Osijek
  - General Hospital Zadar, Zadar
  - Solmed Polyclinic, Zagreb
  - University hospital centre Zagreb, Zagreb
- Czechia (3):
  - Fakultni nemocnice Ostrava, Ostrava
  - Institut klinicke a experimentalni mediciny, Prague
  - Krajska nemocnice T. Bati a.s., Zlín
- France (12):
  - CHU Nice - Hôpital de l'Archet 2, Nice, Alpes Maritimes
  - Hôpital Nord - CHU Marseille, Marseille, Bouches-du-Rhône
  - CHU Caen - Hôpital de la Côte de Nacre, Caen, Calvados
  - Hopital Rangueil, Toulouse, Haute Garonne
  - Institut des MICI, Neuilly, Hauts De Seine
  - CHU Rennes - Hôpital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU de Grenoble - Hôpital Nord, Grenoble, Isere
  - Hospital de brabois, Vantoux, Moselle
  - CHU Lille - Hôpital Claude Huriez, Lille, Nord
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - CHU Amiens - Hopital Sud, Amiens, Somme
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon, Vendée
- Germany (8):
  - Medius Klinik Nuertingen, Nürtingen, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Augsburg, Augsburg, Bavaria
  - INLUGA im Haus der Gesundheit, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Charité - Campus Charité Mitte, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Hamburgisches Forschungsinstitut fure Chronische Darmerkrankungen, Hamburg
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Vasutegeszsegugyi Kft. - Debreceni Egeszsegugyi Kozpont, Debrecen
  - Obudai Egeszsegugyi Centrum Kft., Dunaújváros
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Clinfan Szolgaltato Kft., Szekszárd
- India (16):
  - Origin Hospital, Hyderabad, Andhra Pradesh
  - Yashoda Super Speciality Hospital, Hyderabad, Andhra Pradesh
  - Gandhi Hospital, Secunderabad, Andhra Pradesh
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Gujarat Hospital, Surat, Gujarat
  - Isha Multispeciality Hospital, Vadodara, Gujarat
  - Vinaya Hospital and Research Center, Mangalore, Karnataka
  - Lakeshore Hospital and Research Centre Ltd., Kochi, Kerala
  - Lokmanya Tilak Municipal General Hospital & Medical College, Mumbai, Maharashtra
  - Datta Meghe Institute of Medical Sciences (Deemed University), Wardha, Maharashtra
  - Fortis Escorts Heart Institute and Research Centre, New Delhi, National Capital Territory of Delhi
  - Maharaja Agrasen Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - SRM Institutes for Medical Sciences, Chennai, Tamil Nadu
  - Institute of Post Graduate Medical Education And Research, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education and Research, Chandigarh
- Ireland (5):
  - Midland Regional Hospital, Mullingar, Westmeath
  - Connolly Hospital, Dublin
  - Portiuncula Hospital, Galway
  - University Hospital Galway, Galway
  - Our Lady of Lourdes, Louth
- Israel (9):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center KMC Institute of Gastroenterology and Liver Diseases, Rehovot
- Italy (9):
  - Ospedale di Circolo, Rho, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Università Campus Bio-Medico di Roma, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (44):
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Kokikai Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Iizuka-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Our Lady of the Snow St. Mary's Hospital, Kurume-shi, Fukuoka
  - Kiryu Kosei General Hospital, Kiryu-shi, Gunma
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - NHO Fukuyama Medical Center, Fukuyama-shi, Hiroshima
  - JA-Hiroshima General Hospital, Hatsukaichi-shi, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - NHO Kure Medical Center and Chugoku Cancer Center, Kure-shi, Hiroshima
  - JCHO Hokkaido Hospital, Sapporo, Hokkaido
  - Aoyama Clinic, Kobe, Hyōgo
  - NHO Mito Medical Center, Ibaraki, Ibaraki
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Jiaikai Izuro Imamura Hospital, Kagoshima, Kagoshima-ken
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima, Kagoshima-ken
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Gokeikai Ofuna Chuo Hospital, Kamakura-shi, Kanagawa
  - Kawasaki Municipal Hospital, Kawasaki-shi, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kaiseikai Hattori Clinic, Kumamoto, Kumamoto
  - Mie University Hospital, Tsu, Mie-ken
  - Saiseikai Niigata Hospital, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology, Ōita, Oita Prefecture
  - Okayama University Hospital, Okayama, Okayama-ken
  - NHO Okayama Medical Center, Okayama, Okayama-ken
  - Keiaikai Nakagami Hospital, Okinawa-shi, Okinawa
  - Shinseikai Sai Gastroenterology, Proctology Clinic, Fujiidera, Osaka
  - Kinshukai Infusion Clinic, Osaka, Osaka
  - NHO Osaka National Hospital, Osaka, Osaka
  - JCHO Osaka Hospital, Osaka, Osaka
  - Saga-Ken Medical Centre Koseikan, Saga, Saga-ken
  - Saga University Hospital, Saga, Saga-ken
  - NHO Ureshino Medical Center, Ureshino-shi, Saga-ken
  - Kumagaya General Hospital, Kumagaya-shi, Saitama
  - Matsuaikai Matsuda Hospital, Hamamatsu, Shizuoka
  - Showa University Koto Toyosu Hospital, Kōtoku, Tokyo-To
  - Kitasato University Kitasato Institute Hospital, Minatoku, Tokyo-To
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo-To
- Lithuania (3):
  - Lithuanian University of Health Sciences Kaunas Hospital, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital branch "Seamen's Hospital", Klaipėda
- Mexico (5):
  - Consultorio Medico, InvesclinicMX, Irapuato, Guanajuato
  - Accelerium S de RL de CV, Monterrey, Nuevo León
  - Inspirepharma S. de R.L. de C.V., Monterrey, Nuevo León
  - FAICIC S. de R.L. de C.V., Veracruz
  - Sociedad de Metabolismo y Corazon S.C, Veracruz
- New Zealand (5):
  - Christchurch Hospital NZ, Christchurch
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
- Poland (14):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Trialmed CRS, Kalisz
  - ETG Kielce Zagorska, Kielce
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Centrum Medyczne Plejady, Krakow
  - 1 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ w Lublinie, Lublin
  - ALLMEDICA sp. z o. o., Nowy Targ
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - Medicome Sp. z o.o., Oświęcim
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Nowe zdrowie-CK, Kieltucki i wspolnicy sp. j., Staszów
  - DC-MED, Swidnica
  - Centrum Zdrowia Tuchow Sp. z o.o., Wierzchosławice
- Romania (11):
  - SC Centrul Medical Medicum SRL, Specialitatea Gastroenterologie, Bucharest
  - Spitalul de Oncologie Monza, Bucharest
  - S.C Delta Health Care S.R.L, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - S.C Policlinica CCBR S.R.L, Bucharest
  - Lotus Med SRL, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Centrul Medical Renasterea Craiova, Craiova
  - S.C Pelican Impex S.R.L, Oradea
  - S.C Centrul Medical Valahia S.R.L, Ploieşti
- Serbia (3):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - General Hospital Subotica, Subotica
- Slovakia (10):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - Endomed, s.r.o., Košice
  - Univerzitna nemocnica Martin, Martin
  - KM Management spol. s r.o., Nitra
  - Fakultna nemocnica Nitra, Nitra
  - Gastro I, s.r.o., Prešov
  - Gastro LM s.r.o., Prešov
  - Svet zdravia a.s., Rimavská Sobota
  - Accout Center s.r.o., Šahy
- Spain (10):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, La Coruña
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Centro Medico Teknon, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital General Juan Ramon Jimenez, Huelva
  - Hospital Montecelo, Pontevedra
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Guy's Hospital, London, Greater London